CLINICAL TRIAL: NCT06822972
Title: A Phase II Safety and Efficacy Study of Selinexor in Combination With Bispecific Antibody in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: HCMT/MM2401: Ph2 Study of Selinexor + Bispecific Antibody for RRMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115964
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor + bispecific antibody (Experimental)
  Interventions: Drug: Selinexor 40 mg

INTERVENTIONS:
Drug: Selinexor 40 mg — Patients will receive 40mg of oral SEL, weekly, beginning after they have completed step-up dosing and are 5 (± 2) days out from administration of the first full treatment dose of bispecific antibody therapy for 12 months or until disease progression.

SUMMARY:
The primary objectives of this study are to determine the safety of single agent Selinexor given with commercial bispecific antibody therapy in patients with Relapsed/Refractory Multiple Myeloma (RRMM) and to determine the MRD negativity rate at 10-5 at 12 months post bispecific antibody therapy.

The investigators will enroll 27 patients with RRMM who are receiving commercial bispecific antibody therapy. Patients will be on treatment for 12 months or until disease progression, and will be followed for 24 months. Study assessments include completing a drug diary, having a safety check in call, and have history, clinical assessments, and labs taken.

Twenty-seven patients will provide 80% power in a one-sample chi square test for a proportion assuming that the rate of negative MRD at 10-5 at 12 months post bispecific antibody therapy is 25% in historical control and 50% in the SEL+bispecific antibody experimental treatment group, under a one-sided 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old at the time of informed consent.
2. Willing and able to provide written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
4. A diagnosis of symptomatic multiple myeloma, with relapsed or refractory disease. Patients must have received at least 4 prior lines of therapy. Prior lines of therapy must include a proteasome inhibitor, an immunomodulatory agent, and an CD38 monoclonal antibody, and may include treatment with BCMA antibody conjugates or BCMA directed chimeric antigen receptor (CAR) T cell therapy.
5. All patients must meet criteria for and will receive teclistamab, elranatamab or talquetamab, as per approved label dosing.
6. Patients who have had CRS/ICANS from bispecific antibody must have complete resolution of CRS/ICANS before initiation of SEL
7. Measurable disease as defined by at least one of the following:

   * Serum monoclonal (M) protein ≥1.0 g/dl by protein electrophoresis
   * >200 mg of M protein in the urine on 24 hour electrophoresis
   * Serum immunoglobulin free light chain ≥10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
   * Measurable plasmacytoma
8. Adequate hepatic function measured on labs collected within 28 days of C1D1:

   * Total bilirubin <1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of <3 × ULN), and
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal to <2.5 × ULN.
9. Adequate renal function measured on labs collected within 28 days of C1D1. Adequacy will be determined by creatinine clearance with values of ≥ 15 mL/min meeting inclusion criteria. Creatinine Clearance will be calculated using the Cockcroft and Gault formula [(140 - Age) x Mass (kg)/ (72 x creatinine mg/dL); multiply by 0.85 if female] (Cockcroft 1976).
10. Adequate hematopoietic function measured on labs collected within 7 days of C1D1:

    * Absolute neutrophil count ≥1500/mm3
    * Hemoglobin ≥8.5 g/dL
    * Platelet count ≥100,000/mm3 (patients for whom <50% of bone marrow nucleated cells are plasma cells) or ≥50,000/mm3 (patients for whom ≥50% of bone marrow nucleated cells are plasma cells)
    * Note 1: Patients receiving hematopoietic growth factor support, including erythropoietin, darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), and platelet stimulators (e.g., eltrombopag, romiplostim, interleukin-11) are eligible.
    * Note 2: Patients must have at least a 1-week interval from the last platelet transfusion prior to the Screening platelet assessment. However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study.
11. Patients who are able to become pregnant must have a negative serum pregnancy test at screening.
12. All patients who could become pregnant or could father a child must use highly effective methods of contraception throughout the study and for 5 months following the last dose of study treatment. Highly effective methods of contraception are listed in Section 9.3.1.
13. Female patients must agree not to donate egg during the study treatment period and/or up to 90 days after the last dose of Selinexor. Male patients must agree not to donate sperm during the study treatment period and/or up to 90 days after the last dose of Selinexor.

Exclusion Criteria:

1. Patients who have received and were refractory to selinexor or another specific inhibitor of nuclear exporter (SINE) compound previously. Note: Patients who were exposed to selinexor or another SINE compound but were not refractory are eligible.
2. Patients with any concurrent medical condition or disease (e.g., uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection) that is likely to interfere with study procedures.
3. Patients with any uncontrolled active infection requiring medical or surgical management within 1 week prior to Cycle 1 Day 1 (C1D1). Note: Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are eligible.
4. Females who are pregnant or breastfeeding females.
5. Patients with active, unstable cardiovascular function, as indicated by the presence of any of the following:

   * Symptomatic ischemia
   * Uncontrolled clinically significant conduction abnormalities (e.g., ventricular tachycardia on anti-arrhythmics); note: patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block are eligible
   * Congestive heart failure of New York Heart Association Class ≥3
   * Known left ventricular ejection fraction <40%
   * Myocardial infarction within 3 months prior to C1D1.
6. Patients with well controlled chronic viral hepatitis and/or Human Immunodeficiency Virus can be considered for the study if they meet any of the following conditions:

   * Patients with active hepatitis B virus (Hep B) who have been on antiviral therapy for hepatitis B for >8 weeks and whose viral load is <100 IU/ml prior to first dose of trial treatment
   * Patients with treated or untreated hepatitis C virus (HCV) and successfully treated and "cured" HCV
   * Patients with Human Immunodeficiency Virus (HIV) who have CD4+ T-cell counts ≥ 350 cells/µL and no history of AIDS-defining opportunistic infections in the last year
7. Patients who still have any grade of CRS/ICANS at 5 (± 2) days of administration of the first full treatment dose of bispecific antibody treatment will be excluded
8. Patients with any active gastrointestinal dysfunction interfering with their ability to swallow tablets or any active gastrointestinal dysfunction that could interfere with absorption of study treatment
9. Patients who are unable or unwilling to take supportive medications such as anti-nausea and anti anorexia agents as recommended by the NCCN CPGO for antiemesis and anorexia/cachexia (palliative care)
10. Patients who have any psychiatric, medical, or other condition that, in the opinion of the investigator, could interfere with treatment, compliance, or the ability to give informed consent.
11. Patients with contraindication to any of the required concomitant drugs or supportive treatments
12. Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of selinexor given with commercial bispecific antibody as measured by severity of adverse events | up to 13 months
  Adverse events are defined using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Minimal residual disease (MRD) negativity rate post bispecific antibody therapy | up to 12 months
  MRD at 10^-5 will be performed by Clonoseq (Adaptive Biotechnologies) or, if Clonoseq could not be performed due to inability to obtain/identify original plasma cell clone, by Duke institutional flow cytometry-based MRD assay.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 13 months
  Disease response will be assessed according to the International Myeloma Working Group (IMWG) response criteria
Complete remission (CR) rate | up to 13 months
  Disease response will be assessed according to the International Myeloma Working Group (IMWG) response criteria
Very good partial response (VGPR) rate | up to 13 months
  Disease response will be assessed according to the International Myeloma Working Group (IMWG) response criteria
Partial response (PR) rate | up to 13 months
  Disease response will be assessed according to the International Myeloma Working Group (IMWG) response criteria
Progression free survival (PFS) | up to 13 months
  Disease response will be assessed according to the International Myeloma Working Group (IMWG) response criteria
Number of participants with cytokine release syndrome (CRS) | up to 13 months
  Cytokine release syndrome will be graded according to the Lee criteria for CRS
Grade of cytokine release syndrome (CRS) | up to 13 months
  Cytokine release syndrome will be graded according to the Lee criteria for CRS
Number of participants with immune effector cell associated neurotoxicities (ICANS) | up to 13 months
  Cytokine release syndrome will be graded according to the Lee criteria for CRS
Grade of immune effector cell associated neurotoxicities (ICANS) | up to 13 months
  Cytokine release syndrome will be graded according to the Lee criteria for CRS

CONTACTS AND LOCATIONS:
Overall Officials: Yubin Kang, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No